CLINICAL TRIAL: NCT05311969
Title: Prevalence of Impaired Executive Functions in Institutionalized Elderly
Brief Title: Prevalence of Impaired Executive Functions
Acronym: EXEPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Korian pour le Bien Vieillir (Other)
Collaborators: Gerontopôle des Pays de la Loire (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EXEPA
Record Dates: First submitted 2022-03-11; First posted 2022-04-05 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Executive Dysfunctions
Keywords: executive functions; nursing home; resident; dependence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- groups/cohort (Experimental): participants will perform the various neuropsychological tests provided for in the protocol
  Interventions: Other: cognitive evaluations and non cognitive evaluations

INTERVENTIONS:
Other: cognitive evaluations and non cognitive evaluations — Cognitive evaluations with executive functions evaluations :
  * Mini Mental State Examination
  * Stroop Victoria Test
  * Hayling test
  * Frontal Assessment Battery test mental flexibility:
  * Trial Making Test (TMT) A and B
  * Connection test
  * Alphaflex test
  * Verbal and visuospatial working memory
  * Wechsler Adult Intelligence Scale (WAIS) span
  * Visuo-spatial span
  * Visuo-spatial span simplified version
  * Month Of the Year Backwards (MOTYB) Planning
  * Tinker Toy test
  * Clock Test
  Non-cognitive evaluations:
  The Katz Autonomy Scale Neuropsychiatric Inventory version Care team Geriatric Depression Scale 15-item version Apathy inventory

SUMMARY:
The evaluation of executive functions, as well as the means of stimulating and preserving them, are at the heart of the challenges for maintaining a level of functional autonomy in the elderly, but also during the loss of this functional autonomy and when entering a situation of dependence and/or dementia. Research that has demonstrated the preponderant role of executive functions on functional abilities are examples of this. Components such as planning, organization, initiation, mental flexibility appear to be strongly correlated with the effective performance of complex activities of daily living. In addition, the capacities for autonomy were found to be significantly reduced, and significantly with the severity of the executive deficits. In addition, if these data have since contributed to determining a level of impairment of the executive processes specific to an early loss of autonomy, they are so in the context of early diagnosis of dementia and validation of a detection tool, early loss of autonomy. The scientific advances of the last five years contribute to a better understanding of the impact of executive disorders, but on the other hand, the diversity of the explanatory phenomena of these disorders considerably complicates their nosology within neuro-evolutionary pathologies. Ultimately, an analysis of executive function disorders must take into account cognitive and behavioral aspects, that is to say, beyond performance on tests identified as involving executive functions, behavioral disorders, emotional status and level of autonomy in activities of daily living. In the state of our knowledge, the consideration of executive functions represents a strategic point at the crossroads of the evaluation of the act of care and treatment. Establishing data on the prevalence of alterations in the executive functions of residents, exploring the possibilities of evaluation with a battery of tests little used in this context and linking "executive" profiles and clinical situations seems to us a relevant and interesting first step. However essential to provide a beginning of answer to these questions. This study being an exploratory study. The results of this study will constitute new prevalence data in the population of residents of nursing homes. The aim here is to establish data on the prevalence of alterations in the executive functions of residents, to explore the possibilities of evaluation with a battery of tests little used in this context and to relate the profiles "executives" and clinical situations. This in order to develop a methodology to draw up a general assessment, and to make comparisons of the different profiles, inter/intra pathologies and stages of evolution. Thus, a more in-depth knowledge of the specific profiles of Nursing Home residents will also lead to the reflection of pharmacological and non-pharmacological therapeutic strategies. Finally, it will ultimately be a question of presenting an inventory of the situation of Nursing Home to alert public policies. The main objective is to study the prevalence of impaired executive functions in nursing home residents. The secondary objectives are to explore the feasibility of carrying out executive function tests and to examine the coorelationbetween the levels of impairment of executive functions and the clinical and functional characteristics of residents.

DETAILED DESCRIPTION:
Participants will be recruited by the investigating doctor and the healthcare team. Participants must meet the defined inclusion criteria The steps:

1. Screening Pre-selection of participants potentially eligible for the study (inclusion/non-inclusion criteria) and collection of data from medical records and the healthcare database.

   The information can be collected by the nursing coordinator of the Nursing home. The diagnosis will be determined by the investigating physician of each center and the inclusion criteria checked.
2. Pre-inclusion-inclusion visit

   * Confirmation of eligibility criteria for participants selected for the screening phase
   * Delivery of Consent forms for reading, for explanation of the study methods (procedure, context, objective, constraints), and to answer any questions. If the participant agrees to participate in the study. The consent forms must be signed and dated before any act carried out within the framework of the research. A time of reflection can be granted before the signature. The evaluation of global cognitive functioning with the Mini Mental State Examination will be carried out. Each potentially eligible participant will be given an information note on the conduct of the study followed by an informed consent form that he and the investigator will need to sign before the start of the study.

   The course of the study for the participant will consist of 4 visits with the psychologist and/or the doctor:

   Pre-inclusion consultation, Visit 0: during which the participant will take a questionnaire carried out by the psychologist to assess overall cognitive functioning, and the inclusion consultation by the on-site investigator doctor to check whether the participant corresponds to all study criteria. Following this visit, the participant may choose to participate in the research by signing the consent form.

   The visits will take place as follows, spread over 14 to a maximum of 65 days from Pré-inclusion
3. Visits

Visit 1. (20 to 45 minutes, up to 15 days after Visit 0). This visit will allow to do:

* a clinical assessment with the investigating doctor,
* a behavioral assessment by the nursing staff or the psychologist.
* four cognitive tests for a total duration of approximately 15 minutes carried out by the psychologist.
* Additional visit (10 days later maximum): only if one or more tests have not been carried out or completed during visit 1.

Visit 2. (About 25 minutes, 7 to 10 days after visit Visit 1). This visit will allow you to:

* an evaluation of executive functions by the neuropsychologist with four new cognitive tests:
* Additional visit (10 days later maximum): only if one or more tests have not been carried out or completed during visit 2.

Visit 3. (About 30 minutes, 7 to 10 days after visit Visit 2). This visit will allow you to:

* a final evaluation of executive functions by the neuropsychologist with four new cognitive tests:
* Additional visit (10 days later maximum): only if one or more tests have not been carried out or completed during visit 3.

ELIGIBILITY:
Inclusion Criteria:

* Permanent resident in Nursing Home or in temporary accommodation for more than 3 months
* speak and understand the French language
* Mini Mental State Examination (MMSE) between 7 and 24 dating from 8 maximum days
* Compulsorily affiliated with a social security scheme
* Agree to participate in the study in agreement with the trusted person (if applicable)
* co-signatures of the Consent Form between the investigator and the participant or the person of trust (if applicable)

Exclusion Criteria:

* Refusal to sign the consent form
* Resident in a specialized unit for behavioral disorders (Cognitive Behavioral Unit (CBU), Reinforced Accommodation Unit (RAU), Disoriented Elderly Unit (DEU), Centers of Natural Activities Drawn from Useful Occupations (NADUO) et cetera)
* Communication difficulties, sensory and/or motor deficits
* Medical contraindication in relation to a psychological state that could be altered due to participation in the study
* Resident at end of life (life expectancy < 3 months)
* Resident under legal protection
* Participation within 48 hours prior to inclusion in another research

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of executive functions impairment | 12 months

SECONDARY OUTCOMES:
Rate of passed tests | 12 months
  ability of nursing home residents to pass tests provided for in the protocol to evaluate executive functions
Correlation between executive functions impairment and percentage of dependence residents Correlation between executive functions impairment and percentage of residents with | 12 months
Correlation between executive functions impairment and behavioral disorders | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gilles BERRUT, Study Director — Gerontopôle des Pays de la Loire; Leila LAIFA-MARY, Principal Investigator — Korian; Priscilla CLOT-FAYBESSE, Principal Investigator — Korian
Locations (8):
- France (8):
  - KORIAN La Côte Sauvage, Ars-en-Ré
  - Korian Villa Louisa, Bordeaux
  - Korian Villa Evora, Chartres
  - Korian Le Catelli, L'Huisserie
  - Korian Doubs Rivage, Montbéliard
  - Korian Bois Robillard, Nantes
  - Korian Le Baron, Orléans
  - Korian Les Arcades, Paris

REFERENCES:
- [Background] Miyake A, Friedman NP, Emerson MJ, Witzki AH, Howerter A, Wager TD. The unity and diversity of executive functions and their contributions to complex "Frontal Lobe" tasks: a latent variable analysis. Cogn Psychol. 2000 Aug;41(1):49-100. doi: 10.1006/cogp.1999.0734. PMID 10945922
- [Background] Belleville S, Rouleau N, Van der Linden M. Use of the Hayling task to measure inhibition of prepotent responses in normal aging and Alzheimer's disease. Brain Cogn. 2006 Nov;62(2):113-9. doi: 10.1016/j.bandc.2006.04.006. Epub 2006 Jun 6. PMID 16757076
- [Background] Cummings JL, Mega M, Gray K, Rosenberg-Thompson S, Carusi DA, Gornbein J. The Neuropsychiatric Inventory: comprehensive assessment of psychopathology in dementia. Neurology. 1994 Dec;44(12):2308-14. doi: 10.1212/wnl.44.12.2308. PMID 7991117
- [Background] Dubois B, Slachevsky A, Litvan I, Pillon B. The FAB: a Frontal Assessment Battery at bedside. Neurology. 2000 Dec 12;55(11):1621-6. doi: 10.1212/wnl.55.11.1621. PMID 11113214
- [Background] Fisk JE, Sharp CA. Age-related impairment in executive functioning: updating, inhibition, shifting, and access. J Clin Exp Neuropsychol. 2004 Oct;26(7):874-90. doi: 10.1080/13803390490510680. PMID 15742539
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Makino T, Umegaki H, Suzuki Y, Yanagawa M, Nonogaki Z, Nakashima H, Kuzuya M. Relationship between small cerebral white matter lesions and cognitive function in patients with Alzheimer's disease and amnestic mild cognitive impairment. Geriatr Gerontol Int. 2014 Oct;14(4):819-26. doi: 10.1111/ggi.12176. Epub 2013 Nov 12. PMID 24215176
- [Background] Blanco Martin E, Ugarriza Serrano I, Elcoroaristizabal Martin X, Galdos Alcelay L, Molano Salazar A, Bereincua Gandarias R, Ingles Borda S, Uterga Valiente JM, Indakoetxea Juanbeltz MB, Moraza Lopez J, Barandiaran Amillano M, Fernandez-Martinez M. Dysexecutive syndrome in amnesic mild cognitive impairment: a multicenter study. BMC Neurol. 2016 Jun 4;16:88. doi: 10.1186/s12883-016-0607-2. PMID 27260328
- [Background] Perry RJ, Hodges JR. Differentiating frontal and temporal variant frontotemporal dementia from Alzheimer's disease. Neurology. 2000 Jun 27;54(12):2277-84. doi: 10.1212/wnl.54.12.2277. PMID 10881252
- [Background] Robert PH, Clairet S, Benoit M, Koutaich J, Bertogliati C, Tible O, Caci H, Borg M, Brocker P, Bedoucha P. The apathy inventory: assessment of apathy and awareness in Alzheimer's disease, Parkinson's disease and mild cognitive impairment. Int J Geriatr Psychiatry. 2002 Dec;17(12):1099-105. doi: 10.1002/gps.755. PMID 12461757
- [Background] Roussel M, Lhommee E, Narme P, Czernecki V, Gall DL, Krystkowiak P, Diouf M, Godefroy O; GREFEX study group. Dysexecutive syndrome in Parkinson's disease: the GREFEX study. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2017 Sep;24(5):496-507. doi: 10.1080/13825585.2016.1226248. Epub 2016 Sep 1. PMID 27585478
- [Background] Salthouse TA, Toth J, Daniels K, Parks C, Pak R, Wolbrette M, Hocking KJ. Effects of aging on efficiency of task switching in a variant of the trail making test. Neuropsychology. 2000 Jan;14(1):102-11. PMID 10674802
- [Background] Stuss DT. Functions of the frontal lobes: relation to executive functions. J Int Neuropsychol Soc. 2011 Sep;17(5):759-65. doi: 10.1017/S1355617711000695. Epub 2011 May 24. PMID 21729406
- [Background] Stuss DT, Alexander MP, Shallice T, Picton TW, Binns MA, Macdonald R, Borowiec A, Katz DI. Multiple frontal systems controlling response speed. Neuropsychologia. 2005;43(3):396-417. doi: 10.1016/j.neuropsychologia.2004.06.010. PMID 15707616
- [Background] Tomaszewski Farias S, Cahn-Weiner DA, Harvey DJ, Reed BR, Mungas D, Kramer JH, Chui H. Longitudinal changes in memory and executive functioning are associated with longitudinal change in instrumental activities of daily living in older adults. Clin Neuropsychol. 2009 Apr;23(3):446-61. doi: 10.1080/13854040802360558. Epub 2008 Sep 23. PMID 18821181
- [Background] Torralva T, Roca M, Gleichgerrcht E, Bekinschtein T, Manes F. A neuropsychological battery to detect specific executive and social cognitive impairments in early frontotemporal dementia. Brain. 2009 May;132(Pt 5):1299-309. doi: 10.1093/brain/awp041. Epub 2009 Mar 31. PMID 19336463
- [Background] Torralva T, Roca M, Gleichgerrcht E, Lopez P, Manes F. INECO Frontal Screening (IFS): a brief, sensitive, and specific tool to assess executive functions in dementia. J Int Neuropsychol Soc. 2009 Sep;15(5):777-86. doi: 10.1017/S1355617709990415. Epub 2009 Jul 28. PMID 19635178
- [Background] Tosto G, Zimmerman ME, Hamilton JL, Carmichael OT, Brickman AM; Alzheimer's Disease Neuroimaging Initiative. The effect of white matter hyperintensities on neurodegeneration in mild cognitive impairment. Alzheimers Dement. 2015 Dec;11(12):1510-1519. doi: 10.1016/j.jalz.2015.05.014. Epub 2015 Jun 13. PMID 26079417